CLINICAL TRIAL: NCT02406079
Title: Impact of Tracheotomy on Levels of Serum Procalcitonin in Patients Without Sepsis: a Prospective Study
Brief Title: Impact of Tracheotomy on Procalcitonin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Xingui Dai, First People's Hospital of Chenzhou, First People's Hospital of Chenzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CZ-001
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Tracheotomy
Keywords: tracheotomy; procalcitonin; sepsis
MeSH Terms: conditions — Sepsis | interventions — Tracheotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tracheotomy (Experimental)
  Interventions: Procedure: tracheotomy

INTERVENTIONS:
Procedure: tracheotomy — Tracheotomy is one of most performed surgical procedures to assure airway by making a hole in front of the trachea in ICU.

SUMMARY:
Procalcitonin (PCT) is a reliable biomarker of infection and sepsis. The investigators aimed to determine whether tracheotomy influences PCT concentrations in patients without sepsis, and to assess whether operative duration and procedure affect the peak PCT level.

DETAILED DESCRIPTION:
Procalcitonin (PCT), a soluble protein composed of 116 amino acids with a sequence identical to that of the calcitonin prohormone, has been considered as a reliable biomarker for evaluating of bacterial infection and sepsis. In healthy individuals, serum PCT concentrations are undetectable, however, in case of severe bacterial infections and sepsis, it increase rapidly released mainly in peripheral blood mononuclear cells and modulated by bacterial lipopolysaccharides (LPS) and sepsis-associated cytokines. An increase number of studies have demonstrated that PCT-guided strategy is a helpful approach to guide antibiotic administrations and clinical interventions in the intensive care unit (ICU).

However, PCT is induced in the plasmas of patients not only at the presence of bacterial infection, but also in stress conditions such as severe trauma and surgery. In these conditions, the increases are moderate. The mechanism of the nonspecific increase is complicated. Other conditions with elevated PCT concentrations include medullary thyroid carcinoma , cancer, anaphylactic shock, heat shock , cardiac arrest, Kawasaki Disease, and so on. These findings suggest that elevated PCT levels lack the speciality to detect sepsis in critically ill patients.

Tracheotomy is one of most performed surgical procedures to assure airway by making a hole in front of the trachea in ICU. There are studies in literature that show the surgical procedures to the neck area cause a surgical stress, an increase in thyroid hormones. The procedure may due to miscellaneous clinical signs by altering in hormone levels, even creating a thyroid storm. As far as we are aware, there is no study on the impact of tracheotomy on PCT concentration. The aim of the study was to evaluated whether tracheotomy affects PCT concentrations in patients without sepsis. Moreover, the investigators assessed whether operative duration and procedure were correlation with the peak PCT level.

ELIGIBILITY:
Inclusion Criteria:

* without sepsis requiring tracheotomy

Exclusion Criteria:

* those who did not give their consent or declined treatment during the period of observation
* those with any thyroid diseases past history, such as hyperthyroidism, hypothyroidism and thyroidtumor
* those who received high-dose steroid treatment
* those who received renal replacement therapy (RRT)
* those with severe renal injury (Scr > 300 umol/L)
* those who received antibiotic therapy from 48 hours pre-operation to 72 hours post-operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
procalcitonin | 0-72 hours